CLINICAL TRIAL: NCT00341068
Title: Genetic Analysis of Neural Tube and Orofacial Cleft Defects in the Irish Population
Status: Terminated | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999053; OH99-HG-N053
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12-02

CONDITIONS: Neural Tube Defects (NTDs); Facial Cleft Defect; Hereditary Oral Clefts
Keywords: Birth Defects; Folic Acid; Gene-Environment Interactions; Neural Tube Defects; Cleft Lip
MeSH Terms: conditions — Neural Tube Defects; Congenital Abnormalities; Cleft Lip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Cleft: children and adults with a cleft lip and/or cleft palate and their parents residing in the Republic of Ireland, Northern Ireland and the United Kingdom
- NTD: children and adults with an NTD (neural tube defects) and their parents residing in the Republic of Ireland, Northern Ireland and the United Kingdom

SUMMARY:
In a collaborative effort with the Health Research Board, the national organization for medical research in the Republic of Ireland, individuals with neural tube defects (NTDs) or facial cleft defects and their parents will be studied. With the exception of a few well-described syndromes most cases of NTDs and facial clefts are not inherited in a Mendelian fashion. Nearly all incident cases occur in families with no prior history of the defects. The observed recurrence risk in families with an NTD child is 10-12 fold higher than the general population suggesting that inherited factors modify this risk. Historically, the incidence of NTDs in Ireland was 5-8 fold higher than the USA. The aim of this study is to identify the gene(s) involved in these defects using standard genetic epidemiology approaches, transmission disequilibrium testing and gene mapping strategies. We will initially evaluate genes known to be involved in folate metabolism and pattern formation (development of the body). The major outcomes measured will be aggregate allele frequencies in case groups compared to controls. Biochemical parameters in red cells and plasma will also be measured. Comparisons will be made between the presence of genetics variants, biochemical parameters and clinical phenotype. Characterizing the genes associated with these defects should provide insight into the etiology and metabolic processes that may be involved, furthering prevention and intervention efforts.

DETAILED DESCRIPTION:
In a collaborative effort with the Health Research Board, the national organization for medical research in the Republic of Ireland, individuals with neural tube defects (NTDs) or facial cleft defects and their parents will be studied. With the exception of a few well-described syndromes most cases of NTDs and facial clefts are not inherited in a Mendelian fashion. Nearly all incident cases occur in families with no prior history of the defects. However, the observed recurrence risk in families with an NTD child is 10-20 fold higher than the general population incidence suggesting that inherited factors modify this risk. Historically, the incidence of NTDs in Ireland was 5-8 fold higher than the USA. The aim of this study is to identify the gene(s) involved in these defects using standard genetic epidemiology approaches, transmission disequilibrium testing and gene mapping strategies. We will initially evaluate genes known to be involved in folate metabolism and pattern formation (development of the body). The major outcomes measured will be aggregate allele frequencies in case groups compared to controls. Biochemical parameters in red blood cells and plasma will also be measured. Comparisons will be made between the presence of genetics variants, biochemical parameters and clinical phenotype. Characterizing the genes associated with these defects should provide insight into the etiology and metabolic processes that may be involved, furthering prevention and intervention efforts.

ELIGIBILITY:
* INCLUSION CRITERIA:

Eligible participants are children and adults with an NTD and their parents residing in the Republic of Ireland, Northern Ireland and the United Kingdom

NTDs are defined to include all forms of spina bifida aperta (meningocele, meningomyelocele), encephalocele, anencephaly, rachischisis, iniencephaly and lipomeningocele. Hydrocephalus, hydranencephaly, dermal sinus and spina bifida occulta do not qualify as NTDs.

For oral clefts, eligible participants are children and adults with a facial cleft in Ireland and their parents.

All families with NTDs or clefts will be recruited for the study.

EXCLUSION CRITERIA:

Those with known syndromes will be excluded or analyzed separately.

Cases for whom both biologic parents are not available will be excluded from some components of triad (case, mother and father) analysis, although the data from the NTD case may be useful for other study components.

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7451 (Actual)
Dates: Start 2000-01-01; Study Completion 2019-12-02

PRIMARY OUTCOMES:
Develop list of candidate genes for these disorders | Ongoing
  Develop list of candidate genes for these disorders
Identify intronic and coding polymorphisms in candidate genes | ongoing
  Identify intronic and coding polymorphisms in candidate genes
Score collected samples for association and/or linkage between specific alleles and disease status | ongoing
  Score collected samples for association and/or linkage between specific alleles and disease status

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C Brody, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States